CLINICAL TRIAL: NCT04456075
Title: Risk Prediction and Therapy Monitoring in Patients With SARS-Cov-2 Infection / COVID 19
Acronym: CROWNLESS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Heidelberg University (Other)
Responsible Party: Principal Investigator, Dr. Frederik Trinkmann, Principal Investigator, Heidelberg University
Other Study IDs: CROWNLESS
Record Dates: First submitted 2020-06-29; First posted 2020-07-02 (Actual); Last update posted 2020-07-02 (Actual); Status verified 2020-06

CONDITIONS: SARS-CoV2; COVID

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Approximately 15% of patients with SARS-CoV-2 infection / COVID-19 develop a severe clinical course. This leads to hospitalization and potentially life threatening complications such as pneumonia and respiratory failure. Predictors for early detection and risk stratification are urgently needed. Moreover, only scarce information is available for long-term follow-up and late complications associated with infection. We therefore aimed to find predictors for severe courses of the novel disease as well as to establish strategies for therapeutic monitoring and follow-up.

ELIGIBILITY:
Inclusion Criteria:

* SARS-CoV-2 infection / COVID 19

Exclusion Criteria:

* invasive ventilation
* respiratory failure at admission

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with SARS-CoV-2 infection / COVID 19
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-04-01 (Actual); Primary Completion 2022-04 (Estimated); Study Completion 2022-04 (Estimated)

PRIMARY OUTCOMES:
TLCO | 3-5 days intervals (inpatients)
  Transfer factor for carbon monoxide
TLCO | 1-6 months (outpatients, follow up)
  Transfer factor for carbon monoxide
D5-20 | 3-5 days intervals (inpatients
  frequency dependence of resistance as measured by oscillometry
D5-20 | 1-6 months (outpatients, follow up)
  frequency dependence of resistance as measured by oscillometry
FEV1/FVC | 3-5 days intervals (inpatients)
  forced expiratory volume in 1 s / forced vital capacity (as measured by spirometry)
FEV1/FVC | 1-6 months (outpatients, follow up)
  forced expiratory volume in 1 s / forced vital capacity (as measured by spirometry)

SECONDARY OUTCOMES:
comorbidities | at hospital admission and each follow (every 1-6 months)
  structured questionnaire
clinical symptoms | 3-5 days intervals (inpatients), 1-6 months (outpatients, follow up)
  structured qualitative questionnaire
St. George's Respiratory Questionnaire total score | 3-5 days intervals (inpatients), 1-6 months (outpatients, follow up)
  validated questionnaire (scores range from 0 to 100, with higher scores indicating more limitations)

CONTACTS AND LOCATIONS:
Overall Officials: Frederik Trinkmann, MD, Principal Investigator — Thoraxklinik at Heidelberg University; Felix JF Herth, MD, Study Director — Thoraxklinik at Heidelberg University
Locations (1):
- Thoraxklinik at Heidelberg University, Heidelberg, Germany